CLINICAL TRIAL: NCT00590642
Title: Augment in Treatment-resistent Obsessive-compulsive Disorder: an Open-label Trial
Brief Title: Augmentation in Tx-resistant OCD: an Open Label Trial
Status: Completed | Type: Observational
Sponsor: Creighton University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sriram Ramaswamy, M.D., Creighton University
Other Study IDs: CMP-MD-14
Record Dates: First submitted 2007-12-11; First posted 2008-01-10 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Obsessive Compulsive Disorder
Keywords: obsessive compulsive disorder; OCD; treatment-resistant; SSRI
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
This study examines the use of Acamprosate (Campral(R)) in the treatment of Obsessive Compulsive Disorder (OCD). The treatment of this condition is difficulty and a large percentage of patients fail to respond to medications and have residual symptoms. Such patients are referred to as having treatment resistant OCD.

DETAILED DESCRIPTION:
A patient will receive study drug for about 12 weeks. Throughout the study, the study doctor, on best medical judgment, may gradually increase or decrease the dose of the study medication. The adjustments will dependent on the subject's response and whether the subject has side effects. Once the subject has completed treatment under this study, the subject may resume standard treatment for his/her obsessive compulsive disorder by their regular doctor.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 19-55 years of age
* have dx of OCD as determined by the structured clinical interview for DSM-IV axis 1 disorders
* SSRI resistant patients with OCD
* Subjects who are able to comprehend and satisfactorily comply with protocol requirements and have ability to read and write English.
* Signed written informed consent prior to entering any study procedures.
* Concomitant psychotropic medications permitted only if prescribed at stable dose for at least 1 month before screening visit

Exclusion Criteria:

* Patients with concurrent DSM-IV diagnosis of delirium, dementia, amnestic and other cognitive disorders
* Patients with concurrent DSM-IV diagnosis of mental retardation
* Patients with concurrent DSM-IV diagnosis of lifetime schizophrenia and other psychotic disorders
* Patients with concurrent DSM-IV diagnosis of lifetime bipolar disorder
* Substance dependence or abuse (excluding nicotine) within 6 months prior to screening visit
* Patients with score of less than 16 on Y-BCOS during screening.
* Patients with history of intolerance or hypersensitivity to acamprosate.
* Patients based on history or mental status exam have significant risk fo committing suicide.
* Patients who are homicidal or violent.
* Patients with severe renal impairment
* Female patients who are pregnant or lactating
* Subjects with history of psychosurgery for OCD

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Psychiatry clinic
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Acamprosate would be efficacious for SSRI resistant OCD symptoms | Patients will be administered 12 weeks of Acamprosate.

SECONDARY OUTCOMES:
Acamprosate would improve anxiety, depressive symptoms and quality of life in OCD. | Patients will be administered 12 weeks of Acamprosate

CONTACTS AND LOCATIONS:
Overall Officials: Sriram Ramaswamy, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University Department of Psychiatry, Omaha, Nebraska, United States

REFERENCES:
- [Background] Hollander E, Greenwald S, Neville D, Johnson J, Hornig CD, Weissman MM. Uncomplicated and comorbid obsessive-compulsive disorder in an epidemiologic sample. Depress Anxiety. 1996-1997;4(3):111-9. doi: 10.1002/(SICI)1520-6394(1996)4:33.0.CO;2-J. PMID 9166639
- [Background] Karno M, Golding JM, Sorenson SB, Burnam MA. The epidemiology of obsessive-compulsive disorder in five US communities. Arch Gen Psychiatry. 1988 Dec;45(12):1094-9. doi: 10.1001/archpsyc.1988.01800360042006. PMID 3264144
- [Background] den Boer JA. Psychopharmacology of comorbid obsessive-compulsive disorder and depression. J Clin Psychiatry. 1997;58 Suppl 8:17-9. PMID 9236731
- [Background] Hollander E. Obsessive-compulsive disorder-related disorders: the role of selective serotonergic reuptake inhibitors. Int Clin Psychopharmacol. 1996 Dec;11 Suppl 5:75-87. PMID 9032004
- [Background] Keuneman RJ, Pokos V, Weerasundera R, Castle DJ. Antipsychotic treatment in obsessive-compulsive disorder: a literature review. Aust N Z J Psychiatry. 2005 May;39(5):336-43. doi: 10.1080/j.1440-1614.2005.01591.x. PMID 15860020
- [Background] Saxena S, Rauch SL. Functional neuroimaging and the neuroanatomy of obsessive-compulsive disorder. Psychiatr Clin North Am. 2000 Sep;23(3):563-86. doi: 10.1016/s0193-953x(05)70181-7. PMID 10986728
- [Background] Moore GJ, MacMaster FP, Stewart C, Rosenberg DR. Case study: caudate glutamatergic changes with paroxetine therapy for pediatric obsessive-compulsive disorder. J Am Acad Child Adolesc Psychiatry. 1998 Jun;37(6):663-7. doi: 10.1097/00004583-199806000-00017. PMID 9628087
- [Background] Rosenberg DR, MacMaster FP, Keshavan MS, Fitzgerald KD, Stewart CM, Moore GJ. Decrease in caudate glutamatergic concentrations in pediatric obsessive-compulsive disorder patients taking paroxetine. J Am Acad Child Adolesc Psychiatry. 2000 Sep;39(9):1096-103. doi: 10.1097/00004583-200009000-00008. PMID 10986805
- [Background] Chakrabarty K, Bhattacharyya S, Christopher R, Khanna S. Glutamatergic dysfunction in OCD. Neuropsychopharmacology. 2005 Sep;30(9):1735-40. doi: 10.1038/sj.npp.1300733. PMID 15841109
- [Background] Coric V, Taskiran S, Pittenger C, Wasylink S, Mathalon DH, Valentine G, Saksa J, Wu YT, Gueorguieva R, Sanacora G, Malison RT, Krystal JH. Riluzole augmentation in treatment-resistant obsessive-compulsive disorder: an open-label trial. Biol Psychiatry. 2005 Sep 1;58(5):424-8. doi: 10.1016/j.biopsych.2005.04.043. PMID 15993857
- [Background] Poyurovsky M, Weizman R, Weizman A, Koran L. Memantine for treatment-resistant OCD. Am J Psychiatry. 2005 Nov;162(11):2191-2. doi: 10.1176/appi.ajp.162.11.2191-a. No abstract available. PMID 16263867
- [Background] De Witte P, Littleton J, Parot P, Koob G. Neuroprotective and abstinence-promoting effects of acamprosate: elucidating the mechanism of action. CNS Drugs. 2005;19(6):517-37. doi: 10.2165/00023210-200519060-00004. PMID 15963001
- [Background] Littleton J, Zieglgansberger W. Pharmacological mechanisms of naltrexone and acamprosate in the prevention of relapse in alcohol dependence. Am J Addict. 2003;12(s1):s3-s11. doi: 10.1111/j.1521-0391.2003.tb00492.x. PMID 14972776
- [Background] Dahchour A, De Witte P. Effects of acamprosate on excitatory amino acids during multiple ethanol withdrawal periods. Alcohol Clin Exp Res. 2003 Mar;27(3):465-70. doi: 10.1097/01.ALC.0000056617.68874.18. PMID 12658112
- [Background] Putzke J, Spanagel R, Tolle TR, Zieglgansberger W. The anti-craving drug acamprosate reduces c-fos expression in rats undergoing ethanol withdrawal. Eur J Pharmacol. 1996 Dec 12;317(1):39-48. doi: 10.1016/s0014-2999(96)00696-6. PMID 8982717
- [Background] al Qatari M, Khan S, Harris B, Littleton J. Acamprosate is neuroprotective against glutamate-induced excitotoxicity when enhanced by ethanol withdrawal in neocortical cultures of fetal rat brain. Alcohol Clin Exp Res. 2001 Sep;25(9):1276-83. doi: 10.1097/00000374-200109000-00006. PMID 11584146
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Fleischmann RL, Hill CL, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. I. Development, use, and reliability. Arch Gen Psychiatry. 1989 Nov;46(11):1006-11. doi: 10.1001/archpsyc.1989.01810110048007. PMID 2684084